CLINICAL TRIAL: NCT02888613
Title: Prospective Randomized Study of Two Aortic Surgical Approaches: Mini-laparotomy Versus Mini Lumbotomy
Brief Title: Mini-laparotomy Versus Mini Lumbotomy
Acronym: RAMini
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-A00990-51
Record Dates: First submitted 2016-07-01; First posted 2016-09-05 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Abdominal Aortic Aneurysms; Abdominal Aortic Thrombosis
Keywords: mini-lumbotomy; mini-laparotomy; retroperitoneal approach; transperitoneal approach; abdominal aortic surgery
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini laparotomy (Other): Patients with surgical indication to mini invasive aortic repair will be operated after randomisation with transperitoneal approach
  Interventions: Procedure: mini laparotomy
- Mini lumbotomy (Other): Patients with surgical indication to mini invasive aortic repair will be operated after randomisation with retroperitoneal approach
  Interventions: Procedure: mini lumbotomy

INTERVENTIONS:
Procedure: mini laparotomy — The patient will be positioned supine. After induction of general anesthesia, a median umbilical incision will be performed. The average length of the incision of the laparotomy will be 10 cm (8-12 cm). The small intestine will be then mobilized medially and held by an orthostatic retractor. Arterial dissection and control as well as bypasses will be performed according to the conventional technique. In case of occlusive disease of the iliac arteries, femoral site will be selected to achieve the distal anastomoses of the bifurcated prosthetic graft.
  Other Names: transperitoneal approach
  Arms: Mini laparotomy
Procedure: mini lumbotomy — After induction of general anesthesia, the patient will be positioned in right lateral decubitus at 45° of the table plane. The incision will be performed from the tip of the eleventh rib with a slightly sloping path to the outer edge of the rectus muscle. The average length of the incision of the laparotomy will be 10 cm (8-12 cm).
  Abdominal aorta will be approached retroperitoneally. Arterial dissection and control as well as bypasses will be performed according to the conventional retroperitoneal technique. In case of occlusive disease of the iliac arteries, femoral site will be selected to achieve the distal anastomoses of the bifurcated prosthetic graft.
  Other Names: retro-peritoneal approach
  Arms: Mini lumbotomy

SUMMARY:
This study aims to compare the results of two mini invasive surgical approaches in abdominal aortic surgery: mini lumbotomy with retroperitoneal approach versus mini laparotomy with transperitoneal approach. Respiratory and renal functions and recovery of intestinal transit will be assessed after 30 days.

The secondary purpose of this study is to assess the life quality and morbi-mortality at 30 days, as well as at 6 and 12 months.

DETAILED DESCRIPTION:
Following abdominal aortic surgery, post-operative outcomes are considered favorable with a rapid recovery of respiratory, renal functions and intestinal transit, with limited cardiac events. Complications are still frequent after the classic open abdominal surgery.

In abdominal aortic surgery, "mini" abdominal incision has been proposed as an alternative to the classic large surgical approach.

Two mini surgical approaches are possible: mini lumbotomy with retroperitoneal approach, and mini laparatomy with transperitoneal approach.

Previous studies have only compared classic versus mini surgical approaches and many are retrospectives studies. Pain control through the mini-incision surgery allowed early mobilization of patients, improved lung function, reduced muscle loss, and favoured intestinal motility.

So far, no study has compared the results of two mini invasive aortic approaches.

The aim of this prospective randomized study is to compare two mini-invasive surgical approaches and to determine which of them allows the improvement of surgical outcomes with less morbi-mortality.

ELIGIBILITY:
Inclusion Criteria:

* Elective abdominal aortic repair.
* Abdominal aneurysm or occlusive aortic disease requiring intervention.
* Written consent previously provided by the patient.
* Affiliation to social security.
* Preliminary medical examination.

Exclusion Criteria:

* Hostile abdomen.
* Juxta renal abdominal aortic aneurysm.
* Aneurysmal extension to the iliac arteries.
* Concomitant visceral arteries lesions.
* Urgent surgery.
* Contraindication to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory recovery | day 30
  evaluated with respiratory function test (Sniff nasal inspiratory pressure, SNIP test)
Renal recovery | day 30
  evaluated by blood creatinine level, uremia and kalemia
Intestinal transit recovery | day 30
  evaluated by reapparition of gas and transit

SECONDARY OUTCOMES:
Respiratory recovery | day 1
  evaluated by SNIP test
Respiratory recovery | day 3
  evaluated by SNIP test
Respiratory recovery | day 5
  evaluated by SNIP test
Renal recovery | day 1
  evaluated by creatinine clearance, uremia and kaliemia
Renal recovery | day 3
  evaluated by creatinine clearance, uremia and kaliemia
Renal recovery | day 5
  evaluated by creatinine clearance, uremia and kaliemia
Intestinal recovery | day 1
  assessment of intestinal transit (stool emission)
Intestinal recovery | day 3
  assessment of intestinal transit (stool emission)
Intestinal recovery | day 5
  assessment of intestinal transit (stool emission)
Post-operative pain assessment | day 1
  with VAS scale
Post-operative pain assessment | day 3
  with VAS scale
Post-operative pain assessment | day 5
  with VAS scale
Quality of life assessment | after 6 months
  by using SF-12 questionnaire
Quality of life assessment | after 1 year
  by using SF-12 questionnaire
Morbi-mortality | after 6 months
  evaluated by EQ-5D questionnaire
Morbi-mortality | after 1 year
  evaluated by EQ-5D questionnaire
Morbi-mortality | day 30
  evaluated by non-recovery of functions, eventration and death

CONTACTS AND LOCATIONS:
Overall Officials: Nicla Settembre, MD, PhD, Principal Investigator — Department of vascular and endovascular surgery. Nancy University Hospital

IPD SHARING:
Plan to Share IPD: No